CLINICAL TRIAL: NCT01979978
Title: Healthy Buddies Manitoba: A Cluster Randomized Controlled Effectiveness Trial of Peer Mentoring for Healthy Eights in Children.
Brief Title: Healthy Buddies Manitoba
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H2009:205
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Children; Elementary School Age; Rural and Urban; First Nations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Buddies Curriculum (Experimental): Healthy buddies curriculum delivered by older peers weekly covering three components of healthy living: Physical activity, healthy eating and a healthy body image.
  Interventions: Other: Healthy Buddies Curriculum
- Control (No Intervention): This group received standard school curriculum.

INTERVENTIONS:
Other: Healthy Buddies Curriculum — Each week, intermediate students will receive a 45-minute healthy-living lesson plan from their classroom teacher. Later that week, intermediate students will serve as peer mentors ("Buddies"), teaching a 30-minute lesson to their younger students. The Physical activity (i.e."Go Move!") component of the lesson plans includes 30-minutes of structured aerobic fitness sessions, called fitness loops, with the student pairs twice weekly. The dietary ("Go Fuel!") component includes lessons about distinguishing nutritious and from unhealthy (nutrient poor-energy rich) foods and beverages. The body image ("Go Feel Good!") component, the students are taught to value classmates based on individual traits rather than peer influence.
  Arms: Healthy Buddies Curriculum

SUMMARY:
School-based interventions are generally ineffective for preventing weight gain in children. In 2007, a group from the University of British Columbia, developed a program called Healthy Buddies, that relied on peer mentors to help young children adopt healthy living behaviours. Pilot studies revealed that the program effectively prevented weight gain in children. This trial had never been tested on a large scale using a more scientifically sound study design. We developed a large school-based randomized trial to overcome that limitation and test the hypothesis that that a school-based peer-led healthy living program would reduce adiposity and increase physical activity among children 6-12yrs old.

ELIGIBILITY:
Inclusion Criteria:

* Participating schools need to meet the following eligibility criteria: (1) were within provincial jurisdiction, (2) had a minimum of 200 students per school, (3) offered grades 1 through 6.

Exclusion Criteria:

* Children will be excluded if consent was not received from parents or if they had a condition that limited participation in physical activity.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 647 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Waist circumference | 10 months
  Waist circumference at the top of the iliac crest measured in duplicate with a flexible tape.
BMI-Z score | 10 months
  Body mass index Z score is calculated from weight/height2 and normalized to population normative data for age (months) and sex.

SECONDARY OUTCOMES:
Physical activity | 10 months
  Objectively measured using daily pedometer counts recorded by teachers.
Healthy living knowledge and behaviours | 10 months
  Questionnaires regarding healthy foods and food frequency.
Self efficacy | 10 months
  Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Santos, PhD, Principal Investigator — Healthy Child Manitoba; Jon McGavock, PhD, Study Director — Manitoba Institute of Child Health
Locations (1):
- Manitoba Institute of Child Health - University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Nickel NC, Doupe M, Enns JE, Brownell M, Sarkar J, Chateau D, Burland E, Chartier M, Katz A, Crockett L, Azad MB, McGavock JM, Santos R. Differential effects of a school-based obesity prevention program: A cluster randomized trial. Matern Child Nutr. 2021 Jan;17(1):e13009. doi: 10.1111/mcn.13009. Epub 2020 Aug 20. PMID 32815644
- [Derived] Santos RG, Durksen A, Rabbanni R, Chanoine JP, Lamboo Miln A, Mayer T, McGavock JM. Effectiveness of peer-based healthy living lesson plans on anthropometric measures and physical activity in elementary school students: a cluster randomized trial. JAMA Pediatr. 2014 Apr;168(4):330-7. doi: 10.1001/jamapediatrics.2013.3688. PMID 24515353